CLINICAL TRIAL: NCT05692492
Title: A Randomized, Double-blind, Placebo-controlled Phase 2b Study of ZSP1601 in Adult Subjects With Nonalcoholic Steatohepatitis (NASH)
Brief Title: A Randomized, Double-blind, Placebo-controlled Study of ZSP1601 in Adult Subjects With Nonalcoholic Steatohepatitis (NASH)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZSP1601-22-03
Record Dates: First submitted 2022-12-25; First posted 2023-01-20 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ZSP1601 50mg BID (Experimental)
  Interventions: Drug: ZSP1601
- ZSP1601 100 mg BID (Experimental)
  Interventions: Drug: ZSP1601
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZSP1601 — 50mg BID
  Arms: ZSP1601 50mg BID
Drug: ZSP1601 — 100mg BID
  Arms: ZSP1601 100 mg BID
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this research is to evaluate the efficacy and the safety of two doses of ZSP1601 for 48 weeks versus placebo in adult NASH patients.

ELIGIBILITY:
Inclusion Criteria:

1. NASH histological diagnosis on a liver biopsy performed ≤ 24 weeks before randomization, and NAS≥4 (at least 1 point each in inflammation and ballooning), and fibrosis score F2 or F3, and no other chronic liver disease
2. Subjects having given her/his written informed consent
3. Good compliance with the protocol and agree to have liver biopsy performed
4. Subjects (including their partners) agreed to use effective contraception throughout the study period and up to 24 weeks after discontinuation

Exclusion Criteria:

1. History of cirrhosis or liver biopsy suggestive of cirrhosis
2. Metabolic surgery or new technology treatment for weight loss within 5 years prior to randomization or planned during the study period
3. Type 1 diabetes
4. HIV infection
5. Patients with severe or uncontrollable underlying diseases, unsuitable for treatment with ZSP1601, unable to complete study follow-up, or likely to affect the evaluation of trial results judged by investigator
6. Previous malignancy within 5 years
7. Treatment with hepatoprotective drugs
8. Excessive alcohol consumption for 12 or more consecutive weeks within 1 year prior to screening
9. Pregnant and lactating women or those with a positive serum pregnancy test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-06-03 (Actual); Primary Completion 2026-06-16 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Percent of patients with improvement of steatohepatitis and no worsening of liver fibrosis or improvement in liver fibrosis greater than or equal to one stage and no worsening of the steatohepatitis | 48 weeks
  Percent of patients with improvement of steatohepatitis on overall histopathological reading and no worsening of liver fibrosis on NASH-CRN Fibrosis Score or improvement in liver fibrosis greater than or equal to one stage and no worsening of the steatohepatitis

SECONDARY OUTCOMES:
Percent of patients with resolution of steatohepatitis and no worsening of fibrosis or improvement of fibrosis by at least 1 stage and no worsening of steatohepatitis | 48 weeks
Percent of patients with steatohepatitis improvement and improvement of fibrosis by at least 1 stage | 48 weeks
Percent of patients with steatohepatitis resolution and improvement of fibrosis by at least 1 stage | 48 weeks
Percent of patients with steatohepatitis resolution and no worsening of fibrosis | 48 weeks
Percent of patients with steatohepatitis improvement and no worsening of fibrosis | 48 weeks
Change from baseline in liver fat content (LFC) as measured by MRI-PDFF | 48 weeks
Change from baseline in liver chemistry（ALT,AST,GGT） | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- NanFang Hospital, Guangzhou, China